CLINICAL TRIAL: NCT07395791
Title: Evaluation of the Agreement Between ChatGPT-5 and Anesthesiologists' Predictions and Actual Outcomes in Predicting Postoperative Intensive Care Unit Requirement Based on Preoperative Data
Brief Title: Agreement Between ChatGPT-5 and Anesthesiologists in Predicting Postoperative ICU Requirement
Status: Active, not recruiting | Type: Observational
Sponsor: Beste Mutlu Dağlıoğlu (Other)
Responsible Party: Sponsor-Investigator, Beste Mutlu Dağlıoğlu, Specialist in Anesthesiology and Reanimation, Antalya City Hospital
Organization: Antalya City Hospital (Other)
Other Study IDs: AntalyaCity
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Care
Keywords: Artificial Intelligence; ChatGPT; Anesthesiology; Intensive Care Unit; Postoperative Care; Risk Prediction
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (observational study) — This is a non-interventional observational study. No therapeutic or diagnostic intervention is performed as part of the study.

SUMMARY:
Accurate prediction of postoperative intensive care unit (ICU) requirement is essential for patient safety and efficient use of limited ICU resources. In routine clinical practice, decisions regarding postoperative ICU admission are primarily based on anesthesiologists' preoperative clinical judgment, which may vary among clinicians.

This prospective, observational study aims to evaluate the agreement between predictions made by ChatGPT-5(Chat Generative Pre-trained Transformer) and anesthesiologists regarding postoperative ICU requirement using routinely collected preoperative patient data, and to compare these predictions with actual postoperative ICU admission outcomes.

The study does not involve any intervention, treatment modification, or additional procedures beyond standard clinical care. All patient data are anonymized, and clinical management is not influenced by the model's predictions

DETAILED DESCRIPTION:
Postoperative intensive care unit (ICU) admission is a critical component of perioperative patient management, particularly in patients with increased surgical or anesthetic risk. Accurate preoperative identification of patients who will require postoperative ICU care may improve patient safety and optimize resource allocation.

This study is designed as a prospective, non-interventional observational cohort study conducted in adult patients undergoing elective surgical procedures. Routinely collected preoperative clinical data, including demographic characteristics, comorbidities, laboratory results, and anesthesiologists' assessments, are recorded for each participant.

For each patient, postoperative ICU requirement predictions generated by ChatGPT-5 using structured preoperative data are documented. These predictions are compared with anesthesiologists' preoperative ICU admission assessments and with actual postoperative ICU admission outcomes.

No additional diagnostic or therapeutic interventions are performed as part of the study. Patient care follows standard institutional practice at all times. All collected data are anonymized prior to analysis. Statistical analyses focus on agreement and predictive performance measures, including sensitivity, specificity, and concordance between prediction methods and actual outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Patients undergoing elective surgical procedures requiring preoperative anesthesiology evaluation.
* Availability of complete preoperative clinical data required for postoperative intensive care unit (ICU) need prediction.
* Patients evaluated preoperatively by an anesthesiology specialist.

Exclusion Criteria:

* Patients younger than 18 years of age.
* Emergency surgical procedures.
* Patients with incomplete or missing preoperative clinical data.
* Patients who decline the use of their clinical data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older who underwent elective surgical procedures and received preoperative anesthesiology evaluation at a tertiary care hospital. The study includes patients for whom postoperative intensive care unit (ICU) requirement was assessed based on preoperative clinical data. Patient outcomes were evaluated according to actual postoperative ICU admission status.
Sampling Method: Non-Probability Sample
Enrollment: 938 (Actual)
Dates: Start 2025-12-07 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Agreement Between Predicted and Actual Postoperative ICU Requirement | Within the first 24 hours after surgery
  Agreement between preoperative predictions of postoperative intensive care unit (ICU) requirement made by ChatGPT-5 and anesthesiologists, compared with actual postoperative ICU admission outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Beste Mutlu Dağlıoğlu, Principal Investigator — Antalya City Hospital
Locations (1):
- Antalya City Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided